CLINICAL TRIAL: NCT03404817
Title: Single Dose Crossover Comparative Bioavailability and Food Effect Study of Two EMB-001 Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Embera NeuroTherapeutics, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ERL-PK001; U01DA038879 (NIH)
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Cocaine Use Disorder

STUDY DESIGN:
Intervention Model Description: 3-period, 3-sequence crossover evaluating 3 treatments
  * Treatment-1: new formulation under fed conditions
  * Treatment-2: new formulation under fasted conditions
  * Treatment-3: original formulation under fed conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (Active Comparator): Subjects will receive investigational product (IP) once each Period as a single dose under fasted or fed conditions as follows:
  Period 1: EMB-001 new formulation under fed condition Period 2: EMB-001 new formulation under fasted conditions Period 3: EMB-001 original formulation under fed conditions
  Interventions: Drug: Original formulation EMB-001; Drug: New formulation EMB-001
- Sequence 2 (Active Comparator): Subjects will receive investigational product (IP) once each Period as a single dose under fasted or fed conditions as follows:
  Period 1: EMB-001 original formulation under fed conditions Period 2: EMB-001 new formulation under fed conditions Period 3: EMB-001 new formulation under fasted conditions
  Interventions: Drug: Original formulation EMB-001; Drug: New formulation EMB-001
- Sequence 3 (Active Comparator): Subjects will receive investigational product (IP) once each Period as a single dose under fasted or fed conditions as follows:
  Period 1: EMB-001 new formulation under fasted conditions Period 2: EMB-001 original formulation under fed conditions Period 3: EMB-001 new formulation under fed conditions
  Interventions: Drug: Original formulation EMB-001; Drug: New formulation EMB-001

INTERVENTIONS:
Drug: Original formulation EMB-001 — Single oral dose (720 mg metyrapone/24 mg oxazepam)
Drug: New formulation EMB-001 — Single oral dose (720 mg metyrapone/24 mg oxazepam)

SUMMARY:
This is a study of EMB-001 (a combination of two FDA-approved drugs, metyrapone and oxazepam) in healthy adults.This is a Phase 1, single dose, 3-period, 3-sequence, crossover study in 9 healthy male and female (not of childbearing potential) volunteers. The study will evaluate the bioavailability and food effect of a new formulation of EMB-001 relative to the original formulation of EMB 001.

During the study, a total of 9 eligible subjects will be randomized in a 1:1:1 ratio to each of 3 treatment sequences

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study procedures.
2. Age 18 to 60 and able to read and write English
3. Females must be of non-childbearing potential. Evidence of non-childbearing potential includes documented surgical sterilization (hysterectomy or bilateral oophorectomy) or being postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over age 45 in the absence of other biological or physiological cause. In addition, women must have a documented serum follicle stimulating hormone (FSH) level >40 mIU/mL.
4. Light smokers (<10 cigarettes per day), non-smokers, or ex-smokers
5. Body mass index ≥18.5 and <30 kg/m2
6. Able to take oral medications and willing to adhere to medication regimen during the study
7. No clinically relevant abnormal physical findings at the Screening examination
8. Electrocardiogram without clinically significant abnormality at Screening
9. Normal blood pressure (BP) and heart rate (systolic BP 90 to 140 mmHg; diastolic BP 50 to 90 mmHg; heart rate 50 to 100 beats per minute)
10. No clinically relevant abnormal laboratory findings (general biochemistry, hematology, urinalysis, endocrinology [cortisol]) at Screening
11. Adequate organ function at screening as defined by:

    1. Serum aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN; unless the increased AST is assessed by the Investigator as due to hemolysis and/or hepatic iron deposition); and alanine aminotransferase (ALT) ≤ 2.5 × ULN (unless the increased ALT is assessed by the Investigator as due to hepatic iron deposition).
    2. Normal or elevated levels of serum bilirubin. Serum bilirubin >2× ULN is acceptable if the elevation is attributed to hemolysis with or without Gilbert's syndrome.
    3. Serum creatinine ≤ 1.25 × ULN. If serum creatinine > 1.25 × ULN, then 24-hour measured or calculated (Cockcroft-Gault) glomerular filtration rate ≥ 60 mL/min.
    4. Absolute neutrophil count (ANC) ≥ 1.2 × 109/L.
    5. Platelet count ≥ 100 × 109/L.
    6. Activated partial thromboplastin time (aPTT) and international normalized ratio ≤ 1.25 × ULN, unless the patient is receiving therapeutic anticoagulants.

Exclusion Criteria:

1. Any significant current medical conditions (neurological, cardiovascular [including hypertension], endocrine, thyroid, renal, liver), seizures, delirium or hallucinations, or other unstable medical conditions
2. Known hypersensitivity to or intolerance of oxazepam or metyrapone, or any benzodiazepine
3. Subjects that have confounders of the levels of cortisol and/or cortisol binding globulin, including but not limited to: consuming estrogens, selective estrogen receptor modulators, or herbal/natural estrogen-like compounds; low serum albumin or total protein at screening; history of cirrhosis; hyperthyroidism; other thyroid disease that is untreated and not well-controlled; nephrotic syndrome or other protein-losing enteropathies.
4. Current DSM-5 substance use disorder. Mild tobacco, marijuana, or alcohol use are allowed.
5. Participants who have a positive test result at intake appointment on urine drug screens conducted for illicit drugs, including cannabis.
6. Treatment with an investigational drug or biologic within the 30 days preceding the first dose of study medication or plans to take another investigational drug or biologic within 30 days of study completion (including the follow-up visit)
7. Women of childbearing potential.
8. Have positive serology test results at Screening for human immunodeficiency (HIV) 1/HIV 2 antibodies, Hepatitis B surface antigen (HBsAg) or Hepatitis C Antibody (HCVAb) before Day -2 of this study.
9. Suicidal, homicidal thoughts and behaviors, or evidence of current severe mental illness such as schizophrenia, bipolar disorder or others that may interfere with subject safety or data integrity
10. Use of serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor antidepressants in the 30 days prior to Period 1 or during the study.
11. Use of any prescription, over-the-counter, or herbal medications, vitamins, or mineral supplements within 14 days prior to administration of their first study medication dose

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) of EMB-001 | 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, and 48 hours post drug administration in each Period.
  The AUC0-inf is calculated in a plot of concentration of drug in blood plasma against time and extrapolated to infinity.
Maximum Observed Concentration (Cmax) of EMB-001 | Periods 1-3, pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, and 48 hours post drug administration in each Period.
  Cmax is the maximum observed concentration of drug in blood plasma.
Time to Maximum Concentration (Tmax) of EMB-001 | Periods 1-3, pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, and 48 hours post drug administration in each Period.
  Tmax is the time elapsed from the time of drug administration to maximum plasma concentration.
Apparent Half-Life (t1/2) of EMB-001 | Periods 1-3, pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, and 48 hours post drug administration in each Period.
  Half-life is defined as the time required for the drug plasma concentration to be reduced to half.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 21 days
  Adverse event data (including clinically significant changes in laboratory values) will be compiled for EMB-001.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Detke, MD, Study Director — Embera NeuroTherapeutics, Inc.
Locations (1):
- Collaborative Neuroscience Network, LLC, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No